CLINICAL TRIAL: NCT03049163
Title: Comparison the Topical Anesthesia and Retrobulbar Anesthesia for 27-gauge Vitrectomy for Vitreous Floaters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lin Zhong (Other)
Responsible Party: Sponsor-Investigator, Lin Zhong, Resident, The Eye Hospital of Wenzhou Medical University
Organization: The Eye Hospital of Wenzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYQD131101-01
Record Dates: First submitted 2017-01-28; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Perioperative Pain Experiences
MeSH Terms: interventions — proxymetacaine; methylacetylene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitrectomy under retrobulbar anesthesia (Other): 27-gauge vitrectomy for vitreous floaters under traditional retrobulbar anesthesia
  Interventions: Drug: vitrectomy under topical anesthesia [Proparacaine HCL (Alcaine®)]
- vitrectomy under topical anesthesia (Experimental): 27-gauge vitrectomy for vitreous floaters under topical anesthesia
  Interventions: Drug: vitrectomy under topical anesthesia [Proparacaine HCL (Alcaine®)]

INTERVENTIONS:
Drug: vitrectomy under topical anesthesia [Proparacaine HCL (Alcaine®)] — to observe the anesthesia effect of topical anesthesia of 27-gauge vitrectomy for vitreous floaters
  Other Names: 0.5% proparacaine HCL (Alcaine®, Alcon, TX)

SUMMARY:
Routine anesthesia methods for vitrectomy surgery include retrobulbar and peribulbar anesthesia. However, both methods have potential complications that can vary from minor to severe.

Vitrectomy surgery for vitreous floaters is widely considered straighter forward than other vitreoretinal surgeries.

Hence, the investigators compared the effect of topical anesthesia (with eye drops) and retrobulbar anesthesia for 27-gauge par plana vitrectomy for symptomatic vitreous floaters.

ELIGIBILITY:
Inclusion Criteria:

1. patients who is going to undergo vitrectomy surgery for vitreous floaters
2. age>18 years
3. patients who are willing to participate in this study

Exclusion Criteria:

1. patients who had vitrectomy surgery before
2. patients who had penetrating ocular trauma before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Pain Scale | 2 hour post-operation

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of The Eye Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu RH, Zhang R, Lin Z, Liang QH, Moonasar N. A comparison between topical and retrobulbar anesthesia in 27-gauge vitrectomy for vitreous floaters: a randomized controlled trial. BMC Ophthalmol. 2018 Jul 7;18(1):164. doi: 10.1186/s12886-018-0838-7. PMID 29981573
- [Derived] Lin Z, Zhang R, Liang QH, Lin K, Xiao YS, Moonasar N, Wu RH. Surgical Outcomes of 27-Gauge Pars PLana Vitrectomy for Symptomatic Vitreous Floaters. J Ophthalmol. 2017;2017:5496298. doi: 10.1155/2017/5496298. Epub 2017 Nov 29. PMID 29318039